CLINICAL TRIAL: NCT03313219
Title: Pharmacokinetics and Tolerabilitynce Studies of Gentuximab (Recombinant Anti-VEGFR2 Human-mouse Chimeric Monoclonal Antibody) Injection in the Treatment of Late Recurrence of Metastatic Solid Tumors in China: An Open-label，Non-randomised，Uncontrolled，Dose-escalation，Single Center，Pphase Ia Study in Patients With Late Recurrence of Metastatic Solid Tumors in China
Brief Title: Pharmacokinetics and Tolerancebility Studies of Gentuximab Injection in the Treatment ofPatients With Late Recurrence of Metastatic Solid Tumors in China
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GenSci 043
Record Dates: First submitted 2017-10-06; First posted 2017-10-18 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-10

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gentuximab Injection (Experimental): Patients are assigned to a dose level at the time of study entry and scheduled to receive i.v. of a single dose. The patient enter the subsequent multiple dose i.v. in a 7-day cycle if no DLT in 21 days after the first dose. The study period of each subject will be up to 4 cycles until the tumor progression or unacceptable toxicity. The MTD will be determined by assessing DLT in each cohort from cohort 1 to 6, using a 3+3 dose escalation model. Cohort A begin at 4mg/kg IV and the dose escalated in separate cohorts from 8mg/kg IV, 12mg/kg IV，16mg/kg IV and 20mg/kg IV. If there is no DLT observe in any of these 3 patients in 7 weeks, then the trial proceeds to enroll 3 patients into the next higher dose cohort. If one subject develops a DLT at a specific cohort, an additional 3 patients are enrolled into that same dose cohort. Development of DLTs in more than 1 of 6 patients in a specific dose cohort suggests that the MTD has been exceeded, and further dose escalation is not pursued.
  Interventions: Drug: Gentuximab Injection

INTERVENTIONS:
Drug: Gentuximab Injection — Gentuximab Injection (Recombinant anti-VEGFR2 human-mouse chimeric monoclonal antibody injection)

SUMMARY:
The primary objective is to evaluate the safety and, tolerabilitytolerance, pharmacokinetices and immunogenicity of escalating single doses and subsequent multiple dose of Gentuximab Injection in patients with late recurrence of metastatic solid tumors and to determine the maximum tolerated dose（MTD） and dose limiting toxicities（DLT）.with single and subsequent multiple intravenous infusion in patients with late recurrence of metastatic solid tumors and to provide a basis for the protocol design of later clinical trials.

The secondary objective is to evaluate the pharmacokinetics, pharmacodynamics and immunogenicity, and tumor response of multiple dose of Gentuximab Injection in patients with late recurrence of metastatic solid tumors.

DETAILED DESCRIPTION:
The safety profile of Gentuximab Injection will be explored together with the pharmacokinetics, pharmacodynamics and tumour response to treatment with Gentuximab Injection to recommend the dosing regimen for further clinical studies. The pharmacokinetic properties of Gentuximab Injection will be evaluated after single and multiple dose administrations at different dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Male or female. aged between 18 and 75 years.
* Participants with histopathologically or cytologically diagnosed advanced or metastatic malignant solid tumor.
* Did not respond to standard therapy or no standard therapy is available.
* At least one Measurable lesion.
* At least 4 weeks after the last chemotherapy (at least 14 days from the last medication with oral fluorouracil drugs), at least 6 weeks after the last medication with mitomycin C and nitrosourea; wait for at least a elution periods for 5 half-life if anti-tumor biological products are dosed.
* The subject should restore to ≤1 level (NCI-CTCAE4.03) if they have toxicity response caused by previous treatment, except hair loss.
* Performance status (PS) score, ECOG0-1 level.
* A life expectancy of >3 months.
* Adequate hematologic function, as defined by: Absolute neutrophil count (ANC) ≥1.5×109/L; hemoglobin concentration ≥90g/L (allowing blood transfusion); and platelet count ≥100×109/L.
* Adequate hepatic function, as defined by: ALT ≤ 2.5 × ULN, AST ≤ 2.5 × ULN, TBIL ≤ 1.5 × ULN (liver metastases patients ALT ≤ 5 × ULN, AST ≤ 5 × ULN, TBIL ≤ 3 × ULN).
* Adequate renal function, as defined by: serum creatinine level≤ 1.5 × ULN, creatinine clearance ≥ 60ml / min.
* Adequate coagulation function, as defined by: International normalized ratio (INR) ≤1.5× ULN, activated partial thromboplastin time (aPTT) ≤1.5 x ULN.
* Qualified subjects (male and female) who have fertility must agree to use reliable contraceptive methods (hormones or barriers or abstinence) during the trial and at least 12 weeks after the last administration. Female in childbearing age must be negative for blood pregnancy test within 7 days prior to enrollment.
* Subjects should be informed of the study prior to trial and voluntarily signed a written informed consent.
* The subject is able to communicate well with the investigator and be able to complete the study in accordance with the study.

Exclusion Criteria:

* Subject who has HIV infection, active hepatitis B, hepatitis C or syphilis infection.
* Subject is histologically confirmed as lung squamous cell carcinoma or squamous cell carcinoma of the head and neck, or subjects with lung metastases and metastases with the void ，or bleeding tendency or risk which researchers conformed.
* Has known alcohol or drug dependency.
* Has participated in a clinical study of a non-approved experimental agent within 4 weeks prior to study entry.
* Have serious infection need antibiotic therapy by intravenous injection .
* Has documented and/or symptomatic brain or leptomeningeal metastases.
* Has urinary protein prior to study entry (urinary protein ≥1+，need to detection 24h urinary protein，if 24h urinary protein≥1g,then entry not allowed）.
* Has a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess <6 months before study entry.
* Has a serious or nonhealing wound, ulcer, or bone fracture.
* Has undergone major surgery within 28 days before study entry (not including needle biopsy) or have had significant trauma.
* Has active bleeding within 3 months before enrollment.
* Venous thrombosis currently required treatment; myocardial infarction, stroke, or other severe arterial thromboembolic events occurred within 6 months before enrollment.
* Using anticoagulation and antiplatelet drugs.
* Left ventricular ejection fraction ≤ 50%, New York Heart Association (NYHA) Grade II and above heart failure, uncontroled hypertension (systolic blood pressure> 140 mmHg and/ or diastolic blood pressure> 90 mmHg after treatment with a drug) .
* Is pregnant (confirmed by urine or serum pregnancy test) or lactating.
* Has a known serious allergy reaction to recombination monoclonal antibody (MAb) drug, ,or infusion reaction.
* Is not considered to be suitable for this study, in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-10-11 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | Up to 7 weeks
  Number of Participants With One or More Drug-Related Adverse Events (AEs) or Any Serious Adverse Events (SAEs). A summary of AEs and SAEs considered by the investigator to be drug-related is located in the Reported Adverse Events module. An AE is summarized if the onset date is on or after the first dose of study drug and within 30 days after the last dose, or it occurred before the first dose of study drug and worsened while on the therapy.
Pharmacokinetics: Maximum Concentration (Cmax) in single dose | Cycle 1(day1-day21)& Cycle 2(day 21-day 49): Predose, 15 minute, 3 hours, 6 hours, 12 hours, 24 hours, 48 hours、day 3, day 4, day 7, day 14 after completion of infusion, Cohort 5 only)
Pharmacokinetics: Cmax in multiple dose | Predose and 15 minutes after completion of Infusion at day 21, day 28, day 42，Predose and 15 minutes, 3 hours, 8 hours, 24 hours, 48 hours, 96 hours after completion of Infusion at day 35，Predose at day 49（the last follow-up）
Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) in single dose | Cycle 1(day1-day 21)& Cycle 2(day 21-day49): up to day 21（blood collection time are as follows ：Predose, 15 minutes, 3 hours, 6 hours, 12 hours, 24 hours, 48 hours, day 3, day 4, day 7, day 14 after completion of infusion, Cohort 5 only)
Pharmacokinetics: AUC in multiple dose | From day 21 up to day 49（blood collection time：Predose and 15 minutes after completion of Infusion at day 21, day 28, day 42，Predose and 15 minutes, 3hours, 8hours, 24hours, 48hours, 96hours after completion of Infusion at day 35，Predose at day 49

SECONDARY OUTCOMES:
Adverse Events | 4 weeks after disease progression or 4 weeks after the intolerant toxicity occurs or until the subject begins a new tumor treatment (whichever is shorter)
  Drug-Related Adverse Events (AEs) or Any Serious Adverse Events (SAEs)
Anti-drug antibody:Number of Participants With Anti-drug Antibodies | Cycle 1（day 1-day 21）: Cycle 2:day 21-day 49, cycle 3：day 50-up to study completion, an average of 2 years
  A sample will be considered positive for circulating anti-drug antibodies if it exhibits a post-baseline antibody level that exceeds the upper 95% confidence interval of the mean determined from the normal anti-drug level seen in healthy untreated individuals. A participant will be considered to have an anti-drug response if there are 2 consecutive positive samples or if the final sample tested is positive.
Objective response rate: Number of Participants With Objective Response (ORR) | Time Between Meeting Response Criteria and Progressive Disease or Death Due to Any Cause (Up to 1 year)
  Participants achieved disease control if they had a BOR of CR, PR or SD. Progressive Disease (PD) and those participants which were Not Evaluable (NE) were also reported. According to RECIST v1.1, CR was the disappearance of all non-nodal target lesions, with the short axes of any target lymph node reduced to <10 mm, the disappearance of all nontarget lesions, and the normalization of tumor marker levels (if tumor markers were initially above the upper limit of normal); PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph node), taking as reference the baseline sum diameter. SD was neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD, taking as reference the smallest sum diameter since treatment started.
Progression-free survival (PFS) | Time from randomization to the patient tumor progression or death.（up to 1 year）
  Defined as the time from randomization to the patient tumor progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Principal Investigator — Ethics Committee of Drug Clinical Trials
Locations (1):
- Shanghai East Hospital, Shanghai, China